CLINICAL TRIAL: NCT04219332
Title: Comparison of Submucosal and Subserosal Approaches Toward Optimized Indocyanine Green Tracer-Guided Laparoscopic Lymphadenectomy for Patients With Gastric Cancer: The FUGES-019 Randomized Clinical Trial
Brief Title: Randomized Controlled Trial on Effect of Lymph Node Mapping by Indocyanine Green Via Submucosal or Subserosal Injection
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Director, Head of Department of Gastric Surgery, Principal Investigator, Clinical Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FUGES-019
Record Dates: First submitted 2020-01-01; First posted 2020-01-07 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Indocyanine Green; Gastric Cancer; Injection Site
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Although it was not feasible to blind the surgeons and participants, the pathologists were unaware of the intervention received by the patients. The researcher performing the statistical analyses was blinded to the patient group allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Subserosal injection of indocyanine green tracer group (Experimental): Subserosal injection of indocyanine green, with a concentration of 0.5 mg /ml, 6 points along the lesser and greater curvature of the stomach, 1.5 ml for each point.
  Interventions: Drug: Subserosa injection of indocyanine green
- Submucosal injection of indocyanine green tracer group (Active Comparator): Submucosal injection of indocyanine green, with a concentration of 1.25mg /ml, four points around the primary tumor, each point 0.5 ml.
  Interventions: Drug: submucosal injection of indocyanine green

INTERVENTIONS:
Drug: Subserosa injection of indocyanine green — After preoperative exploration, the indocyanine green powder (Dandong Yichuang Pharmaceutical Co) is dissolved in 0.5 mg/ml of sterile water and the prepared solution (1.5 ml for each point) is injected along the subserosal of the stomach at 6 specific points along the lesser and greater curvature of the stomach.
  Other Names: No other intervention
  Arms: Subserosal injection of indocyanine green tracer group
Drug: submucosal injection of indocyanine green — One day before surgery, 1.25 mg/ml indocyanine green (Dandong Yichuang Pharmaceutical Co) was prepared in sterile water and 0.5 ml of the solution was injected into the submucosal layer at 4 quadrants around the primary tumor, amounting to 2.5 mg of indocyanine green.
  Other Names: No other intervention
  Arms: Submucosal injection of indocyanine green tracer group

SUMMARY:
The purpose of this study was to evaluate whether submucosal or subserous injection of indocyanine green during laparoscopic lymphadenectomy for patients with gastric cancer was different. The patients with gastric adenocarcinoma (cT1-4a, N0/+, M0) were studied.

DETAILED DESCRIPTION:
In recent years, with the successful application of ICG (indocyanine green) fluorescence imaging technology in laparoscopic equipment, scholars have found that ICG near-infrared imaging has better tissue penetration and can better identify lymph nodes in hypertrophic adipose tissue than other dyes under visible light, which makes ICG fluorescence imaging guide laparoscopic radical resection of gastric cancer lymph node dissection has become a new exploration direction. ICG near-infrared imaging technology has important research value, good application prospects, and broad development space in laparoscopic radical resection of gastric cancer. However, at present, the application of ICG near-infrared imaging technology in laparoscopic radical resection of gastric cancer is still in the exploratory stage, and there is no unified standard. Therefore, in the world, there is still a lack of high-level evidence-based evidence of large-sample prospective randomized controlled trials to evaluate the effectiveness, safety, and feasibility of submucosal or subserous injection of ICG in guiding laparoscopic D2 resection of gastric cancer. The investigator first carried out this study in the world to evaluate the lymph node dissection and perioperative safety of gastric cancer patients who received a submucosal injection of ICG and subserous injection of ICG during laparoscopic radical gastrectomy in the same period, to promote the standardized development of ICG near-infrared imaging in laparoscopic radical gastrectomy.

ELIGIBILITY:
Inclusion criteria:

1. Age from 18 to 75 years
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. Clinical stage tumor T1-4a (cT1-4a), N0/+, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Eighth Edition. Preoperative staging was made by conducting mandatory computed tomography (CT) scans and an optional endoscopic ultrasound
4. No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative examinations
5. Performance status of 0 or 1 on Eastern Cooperative Oncology Group scale (ECOG)
6. American Society of Anesthesiology score (ASA) class I, II, or III
7. Written informed consent

Exclusion criteria:

1. Women during pregnancy or breast-feeding
2. Severe mental disorder
3. History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
4. History of previous gastrectomy, endoscopic mucosal resection or endoscopic submucosal dissection
5. Rejection of laparoscopic resection
6. History of allergy to iodine agents
7. Enlarged or bulky regional lymph node diameter over 3cm by preoperative imaging
8. History of other malignant disease within past five years
9. History of previous neoadjuvant chemotherapy or radiotherapy
10. History of unstable angina or myocardial infarction within past six months
11. History of cerebrovascular accident within past six months
12. History of continuous systematic administration of corticosteroids within one month
13. Requirement of simultaneous surgery for other disease
14. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
15. Forced expiratory volume in 1 second (FEV1)<50% of predicted values
16. Linitis plastica, Widespread

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2019-12-31 (Actual); Primary Completion 2020-11-27 (Actual); Study Completion 2023-10-28 (Estimated)

PRIMARY OUTCOMES:
Total Number of Retrieved Lymph Nodes | One month after surgery
  Total Number of Retrieved Lymph Nodes

SECONDARY OUTCOMES:
Total number of fluorescent lymph nodes in groups A and B | One month after surgery
  Total number of fluorescent lymph nodes in groups A and B
Relationship between fluorescent lymph nodes and positive lymph nodes in groups A and B (true positive rate) | One month after surgery
  Relationship between fluorescent lymph nodes and positive lymph nodes in groups A and B (true positive rate)
Relationship between fluorescent lymph nodes and negative lymph nodes in groups A and B (false positive rate) | One month after surgery
  Relationship between fluorescent lymph nodes and negative lymph nodes in groups A and B (false positive rate)
Relationship between non-fluorescent and negative lymph nodes in groups A and B (true negative rate) | One month after surgery
  Relationship between non-fluorescent and negative lymph nodes in groups A and B (true negative rate)
Relationship between non-fluorescent lymph nodes and positive lymph nodes in groups A and B (false negative rate) | One month after surgery
  Relationship between non-fluorescent lymph nodes and positive lymph nodes in groups A and B (false negative rate)
Number of Metastasis Lymph Nodes | One month after surgery
  Number of Metastasis Lymph Nodes
Metastasis rate of lymph node | One month after surgery
  Metastasis rate of lymph node
Mortality rates | 30 days
  This is for the early mortality, which defined as the event observed within 30 days after surgery.
Morbidity rates | 30 days
  This is for the incidence of early postoperative complications, which defined as the event observed within 30 days after surgery.
3-year disease free survival rate | 36 months
  Disease-free survival is calculated from the day of surgery to the day of recurrence or death (When the specific date of recurrence of the tumor is unknown, the endpoint is the date of death due to tumor causes). If neither death nor recurrence of the tumor is observed, the endpoint is the final date that a patient is confirmed as relapse-free. (The final date of DFS: The last date of the outpatient visit day or the date of acceptance of the examination).
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
The variation of weight | 3, 6, 9 and 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The variation of BMI in kg/m^2 | 3, 6, 9 and 12 months
  The variation of BMI in kg/m^2 on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
Intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
The variation of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of hemoglobin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein IN milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
Lymph node noncompliance rate | 1 day
  Lymph node noncompliance was defined as the absence of lymph nodes that should have been excised from more than 1 lymph node station. Major lymph node noncompliance was defined as more than 2 intended lymph node stations that were not removed.
Modified EORTC cancer in-patient satisfaction with care measure (EORTC IN-PATSAT14) | 30 days
  Participants were asked to complete one modified European Organisation for Research and Treatment of Cancer (EORTC) IN-PATSAT14 questionnaire before their discharge from hospital.
The Surgery Task Load Index (SURG-TLX) | 1 day
  Surgeons were required to complete one modified SURG-TLX questionnaire for each procedure.
3-year overall survival rate | 36 months
  The overall survival is calculated from the day of surgery until death or until the final follow-up date, whichever occurs first. For survival cases, the endpoint is the last date that survival was confirmed. If the loss to follow-up occurred, the endpoint is the final date that survival could be confirmed.

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ming Huang, MD, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Department of Gastric Surgery, Fuzhou, Fujian, China

REFERENCES:
- [Background] Lee JH, Ryu KW, Kim CG, Kim SK, Choi IJ, Kim YW, Chang HJ, Bae JM, Hong EK. Comparative study of the subserosal versus submucosal dye injection method for sentinel node biopsy in gastric cancer. Eur J Surg Oncol. 2005 Nov;31(9):965-8. doi: 10.1016/j.ejso.2005.03.006. PMID 15908163
- [Background] Kwon IG, Son T, Kim HI, Hyung WJ. Fluorescent Lymphography-Guided Lymphadenectomy During Robotic Radical Gastrectomy for Gastric Cancer. JAMA Surg. 2019 Feb 1;154(2):150-158. doi: 10.1001/jamasurg.2018.4267. PMID 30427990
- [Background] Cianchi F, Indennitate G, Paoli B, Ortolani M, Lami G, Manetti N, Tarantino O, Messeri S, Foppa C, Badii B, Novelli L, Skalamera I, Nelli T, Coratti F, Perigli G, Staderini F. The Clinical Value of Fluorescent Lymphography with Indocyanine Green During Robotic Surgery for Gastric Cancer: a Matched Cohort Study. J Gastrointest Surg. 2020 Oct;24(10):2197-2203. doi: 10.1007/s11605-019-04382-y. Epub 2019 Sep 4. PMID 31485904
- [Background] Herrera-Almario G, Patane M, Sarkaria I, Strong VE. Initial report of near-infrared fluorescence imaging as an intraoperative adjunct for lymph node harvesting during robot-assisted laparoscopic gastrectomy. J Surg Oncol. 2016 Jun;113(7):768-70. doi: 10.1002/jso.24226. Epub 2016 Mar 29. PMID 27021142
- [Background] Chen QY, Zhong Q, Liu ZY, Xie JW, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Tu RH, Huang ZN, Lin JL, Li P, Zheng CH, Huang CM. Does Noncompliance in Lymph Node Dissection Affect Oncological Efficacy in Gastric Cancer Patients Undergoing Radical Gastrectomy? Ann Surg Oncol. 2019 Jun;26(6):1759-1771. doi: 10.1245/s10434-019-07217-x. Epub 2019 Feb 12. PMID 30756329
- [Background] Bredart A, Bottomley A, Blazeby JM, Conroy T, Coens C, D'Haese S, Chie WC, Hammerlid E, Arraras JI, Efficace F, Rodary C, Schraub S, Costantini M, Costantini A, Joly F, Sezer O, Razavi D, Mehlitz M, Bielska-Lasota M, Aaronson NK; European Organisation for Research and Treatment of Cancer Quality of Life Group and Quality of Life Unit. An international prospective study of the EORTC cancer in-patient satisfaction with care measure (EORTC IN-PATSAT32). Eur J Cancer. 2005 Sep;41(14):2120-31. doi: 10.1016/j.ejca.2005.04.041. PMID 16182120
- [Background] Wilson MR, Poolton JM, Malhotra N, Ngo K, Bright E, Masters RS. Development and validation of a surgical workload measure: the surgery task load index (SURG-TLX). World J Surg. 2011 Sep;35(9):1961-9. doi: 10.1007/s00268-011-1141-4. PMID 21597890
- [Background] Tajima Y, Yamazaki K, Masuda Y, Kato M, Yasuda D, Aoki T, Kato T, Murakami M, Miwa M, Kusano M. Sentinel node mapping guided by indocyanine green fluorescence imaging in gastric cancer. Ann Surg. 2009 Jan;249(1):58-62. doi: 10.1097/SLA.0b013e3181927267. PMID 19106676
- [Background] Chen QY, Xie JW, Zhong Q, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Tu RH, Huang ZN, Lin JL, Zheng HL, Li P, Zheng CH, Huang CM. Safety and Efficacy of Indocyanine Green Tracer-Guided Lymph Node Dissection During Laparoscopic Radical Gastrectomy in Patients With Gastric Cancer: A Randomized Clinical Trial. JAMA Surg. 2020 Apr 1;155(4):300-311. doi: 10.1001/jamasurg.2019.6033. PMID 32101269
- [Derived] Chen QY, Zhong Q, Li P, Xie JW, Liu ZY, Huang XB, Lin GT, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Zheng QL, Tu RH, Huang ZN, Zheng CH, Huang CM. Comparison of submucosal and subserosal approaches toward optimized indocyanine green tracer-guided laparoscopic lymphadenectomy for patients with gastric cancer (FUGES-019): a randomized controlled trial. BMC Med. 2021 Oct 27;19(1):276. doi: 10.1186/s12916-021-02125-y. PMID 34702260

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-09-30): https://cdn.clinicaltrials.gov/large-docs/32/NCT04219332/Prot_SAP_ICF_000.pdf